CLINICAL TRIAL: NCT01331564
Title: Electronically-Mediated Weight Interventions for Pregnant and Postpartum Women
Brief Title: eMOMS of Rochester
Acronym: eMOMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Cornell University (Other)
Responsible Party: Principal Investigator, Diana Fernandez, Associate Professor of Public Health Sciences, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HL096760
Record Dates: First submitted 2011-03-31; First posted 2011-04-08 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Gestational Weight Gain; Postpartum Weight Retention
Keywords: Pregnancy; Postpartum; Weight gain; Weight retention; Behavior; Electronic Media; Randomized Clinical Trial
MeSH Terms: conditions — Gestational Weight Gain; Weight Gain; Behavior | interventions — Postpartum Period; Pregnancy; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- electronic intervention group 2 (Experimental): (e-intervention 2) receives a behavioral intervention through a website during pregnancy and until 18 months postpartum
  Interventions: Behavioral: electronic intervention during pregnancy and postpartum
- electronic intervention group 1 (Experimental): (e-intervention 1) receives a behavioral intervention through a website during pregnancy. During the postpartum period this arm receives the same non-weight-related information as the control arm
  Interventions: Behavioral: electronic intervention during pregnancy
- Control (Placebo Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: electronic intervention during pregnancy and postpartum — Electronically-mediated behavioral interventions to encourage women to gain an appropriate amount of weight during pregnancy and to follow a healthy lifestyle postpartum to minimize postpartum weight retention
  Other Names: Behavior modification intervention for pregnancy; Behavior modification intervention for postpartum; Prevention of excessive gestational weight gain; Prevention of postpartum weight retention; Electronically-mediated behavioral interventions
  Arms: electronic intervention group 2
Behavioral: electronic intervention during pregnancy — Electronically-mediated behavioral interventions to encourage women to gain an appropriate amount of weight during pregnancy.
  Other Names: Behavior modification intervention for pregnancy; Prevention of excessive gestational weight gain; Electronically-mediated behavioral interventions
  Arms: electronic intervention group 1
Behavioral: Control — Control women will receive non-weight related content during both time periods at the project website.
  Other Names: Control group
  Arms: Control

SUMMARY:
The project aims to develop, implement and evaluate electronically-mediated behavioral intervention programs for pregnant and postpartum women in order to prevent excessive weight gain during pregnancy and postpartum weight retention.

DETAILED DESCRIPTION:
This study seeks to expand the understanding of how to slow the accumulation of weight in childbearing women. The intervention goals are to decrease the prevalence of excessive pregnancy weight gain and mean weight retention in the first 18 months postpartum in socio-economically and racially/ethnically diverse sample of 1,641 pregnant women. Women will be randomly assigned to one of three groups: Intervention Group 1 will receive the intervention program only during pregnancy (e-intervention 1). Intervention Group 2 will receive e-intervention 1 plus intervention for 18 months postpartum (e-intervention 2). Control women will receive non-weight related content during both time periods at the project website. The primary hypotheses for the randomized controlled trial are: H1: The proportion of women in Intervention Groups 1 and 2 who gain more weight in pregnancy than is recommended by the IOM will be 33% less than the proportion of the women in the Control Group who gain excessively and H2: The Control Group will have a higher mean weight retention at 12 months postpartum than Intervention Groups 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 35 at the time of delivery
* Consented at or before 20 weeks gestation
* Intending to be available for a 24 months intervention
* Plan to deliver in one of the 4 hospitals in Rochester, NY (the study area)
* Plan to carry the pregnancy to term
* Plan to keep the baby
* Read and understand English

Exclusion Criteria:

* BMI < 18.5 kg/m2 and > 35.0 kg/m2.
* Multiple gestation. If multiple gestation is diagnosed after enrollment participant will be terminated from the study (reasons for termination will be included in the consent form)
* Medical conditions prior to pregnancy which could influence weight loss or gain: cystic fibrosis, hyperthyroidism, renal insufficiency1, proteinuria1, cerebral palsy, lupus erythematosus; rheumatoid arthritis, Crohns disease (severity and other autoimmune diseases evaluated case by case), ulcerative colitis, maternal congenital heart disease (patients are often underweight); hypertension treated with medication2,
* Psychiatric medication associated with major weight gain or loss (e.g.; Lithium & Divalproex) Common Criteria
* Household member on study staff
* Past or planned (within the next 24 months) weight loss surgery (e.g. gastric bypass, lap band, or liposuction); current participation in a commercial weight loss program (e.g. Weight Watcher's, Jenny Craig); currently enrolled or planned to enroll in a weight loss or another weight gain prevention study
* Participants will be excluded during screening if they report regular use of systemic steroids, prescription weight loss drugs, and/or diabetes medications (oral or injected- insulin, metformin, byetta, TZDs, other). "Regular use" is defined as "taking this medication most days of the week for the previous month"
* Current treatment for eating disorder
* Positive screening for bulimia
* Weight loss of more than 15 pounds in the three months prior to pregnancy
* Cardiovascular event (heart attack, stroke, episode of heart failure, or revascularization procedure) within the last 6 month. Revascularization is defined as bypass surgery or stints
* Mental or psychiatric condition that precludes giving informed consent and completing questionnaires
* Current treatment for malignancy (other than non-melanoma skin cancer and CIN cervix) or on remission for less than 5 years
* Blood pressure criterion

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1641 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of women whose gestational gain is within the recommended gestational weight gain Institute of Medicine Guidelines in kilograms | 40 weeks
  Gestational weight gain is the result of the last predelivery weight minus the prepregnancy weight (or early pregnancy weight).
Postpartum weight retention in kg at 12 months postpartum | 1.5 years
  The difference between the weight at 12 months postpartum and the pre-pregnancy weight (or early pregnancy weight. Participants will be followed for a maximum of 2 years from recruitment in early pregnancy to 18 months postpartum. The final outcome in the postpartum period is postpartum weight retention at 18 months. Interim measure of postpartum weight will be collected at 6 and 12 months for analyses. The primary hypothesis for the postpartum period is weight retention at 12 months postpartum.

SECONDARY OUTCOMES:
Caloric Intake in Kilocalories | 2 years
  Caloric intake will be calculated based on the average food intake assessed by 2 24-hour dietary recall.
Physical activity as an average weekly energy expenditure (METS) | 2 years
  Physical activity during pregnancy is measured using the Pregnancy Physical Activity Questionnaire and during postpartum using the Global Physical Activity Questionnaire.
Postpartum weight retention at 18 months | 2 years
  The difference between the weight at 18 months postpartum and the prepregnancy weight (or early pregnancy weight). Participants will be followed for a maximum of 2 years from recruitment in early pregnancy to 18 months postpartum. The final outcome in the postpartum period is postpartum weight retention at 18 months. Interim measure of postpartum weight will be collected at 6 and 12 months for analyses. The primary hypothesis for the postpartum period is weight retention at 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Isabel D Fernandez, MD, MPH, PhD, Principal Investigator — University of Rochester; Christine M Olson, PhD, Principal Investigator — Cornell University
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Yu Y, Ma Q, Fernandez ID, Groth SW. Mental Health, Behavior Change Skills, and Eating Behaviors in Postpartum Women. West J Nurs Res. 2022 Oct;44(10):932-945. doi: 10.1177/01939459211021625. Epub 2021 Jun 4. PMID 34088249
- [Derived] Olson CM, Groth SW, Graham ML, Reschke JE, Strawderman MS, Fernandez ID. The effectiveness of an online intervention in preventing excessive gestational weight gain: the e-moms roc randomized controlled trial. BMC Pregnancy Childbirth. 2018 May 9;18(1):148. doi: 10.1186/s12884-018-1767-4. PMID 29743026
- [Derived] Olson CM, Strawderman MS, Graham ML. Association between consistent weight gain tracking and gestational weight gain: Secondary analysis of a randomized trial. Obesity (Silver Spring). 2017 Jul;25(7):1217-1227. doi: 10.1002/oby.21873. Epub 2017 Jun 2. PMID 28573669
- [Derived] Graham ML, Strawderman MS, Demment M, Olson CM. Does Usage of an eHealth Intervention Reduce the Risk of Excessive Gestational Weight Gain? Secondary Analysis From a Randomized Controlled Trial. J Med Internet Res. 2017 Jan 9;19(1):e6. doi: 10.2196/jmir.6644. PMID 28069560
- [Derived] Fernandez ID, Groth SW, Reschke JE, Graham ML, Strawderman M, Olson CM. eMoms: Electronically-mediated weight interventions for pregnant and postpartum women. Study design and baseline characteristics. Contemp Clin Trials. 2015 Jul;43:63-74. doi: 10.1016/j.cct.2015.04.013. Epub 2015 May 6. PMID 25957183
- [Derived] Demment MM, Graham ML, Olson CM. How an online intervention to prevent excessive gestational weight gain is used and by whom: a randomized controlled process evaluation. J Med Internet Res. 2014 Aug 20;16(8):e194. doi: 10.2196/jmir.3483. PMID 25143156